CLINICAL TRIAL: NCT01652261
Title: Very Early FDG-PET/CT-response Adapted Therapy for Advanced Stage Hodgkin Lymphoma, a Randomized Phase III Non-inferiority Study of the EORTC Lymphoma Group
Brief Title: Very Early FDG-PET/CT-response Adapted Therapy for Advanced Hodgkin Lymphoma (H11)
Acronym: H11
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study closed due to lack of recruitment
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Polish Lymphoma Research Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-20101-23101; 2011-005473-22 (EudraCT Number)
Record Dates: First submitted 2012-07-18; First posted 2012-07-30 (Estimated); Last update posted 2021-02-15 (Actual); Status verified 2014-06

CONDITIONS: Hodgkin Lymphoma
Keywords: advanced stage
MeSH Terms: conditions — Hodgkin Disease | interventions — ABVD protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- experimental arm (Experimental): An experimental arm (early FDG-PET/CT-response adapted), where all patients are initially treated with a single cycle of ABVD. Very early FDG-PET/CT-negative patients continue on ABVD therapy to a total of six cycles. Very early FDG-PET/CT-positive patients receive 3 cycles of BEACOPPesc followed by another 3 cycles of BEACOPPesc. Mid-treatment evaluation is performed after 4 cycles. In case of treatment failure (less than partial remission (PR)), the patient goes off protocol treatment.
  Only patients with residual FDG-PET/CT-positive disease after chemotherapy will receive radiotherapy (36 Gy/18 fractions on the FDG-PET/CT-positive residual mass(es)).
  Interventions: Drug: ABVD + FDG-PET/CT Scan treatment adaptation; Drug: BEACOPPesc
- standard arm (Active Comparator): A standard arm, where patients are treated with four cycles of BEACOPPesc followed by 2 cycles of BEACOPPesc. FDG-PET/CT is performed after one cycle, but with no therapeutic consequences. Mid-treatment evaluation is performed after four cycles. In case of treatment failure (less than PR), the patient goes off protocol treatment.
  Only patients with residual FDG-PET/CT-positive disease after chemotherapy will receive radiotherapy (36 Gy/18 fractions on the FDG-PET/CT-positive residual mass(es)).
  Interventions: Drug: BEACOPPesc

INTERVENTIONS:
Drug: ABVD + FDG-PET/CT Scan treatment adaptation
  Arms: experimental arm
Drug: BEACOPPesc

SUMMARY:
The main objective of the trial is to show that doxorubicin, bleomycin, vinblastine, and dacarbazine (ABVD)-based response-adapted therapy for advanced-stage Hodgkin lymphoma, with treatment intensification (bleomycin, etoposide, adriamycin, cyclophosphamide, vincristine, procarbazine, and prednisone (BEACOPPesc) in case of a positive fluorodeoxyglucose (FDG) positron emission tomography (PET) computed tomography (CT) after one cycle of ABVD, has non-inferior efficacy compared with the intensive BEACOPPesc regimen. A second objective is to assess the prognostic value of FDG-PET/CT after one cycle of BEACOPPesc.

ELIGIBILITY:
Inclusion criteria:

* Previously untreated, histologically proven classical Hodgkin lymphoma
* Clinical stages III/IV (Ann Arbor)
* Age 18-60
* WHO performance 0-2
* Adequate organ function
* Patients of childbearing/reproductive potential should use adequate birth control measures during the whole duration of study treatment.
* Written informed consent according to ICH/EU Good Clinical Practice, and national/local regulations

Exclusion criteria:

* Pregnancy or lactation
* Specific contraindications to BEACOPPesc therapy, including:
* Poorly controlled diabetes mellitus
* HIV infection,
* Chronic active hepatitis B and/or hepatitis C
* Concomitant or previous malignancies with the exception of basal cell skin tumors, adequately treated carcinoma in situ of the cervix and any cancer that has been in complete remission for >5 years
* Psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Freedom from treatment failure | 9 years after first patient in (FPI)

SECONDARY OUTCOMES:
response at the end of therapy | 9 years after FPI
Progression-free survival | 9 years after FPI
Overall survival | 9 years after FPI
Acute toxicity | 9 years after FPI
  * Hematological toxicity (blood cell count) can be significant especially for patients who will receive BEACOPPesc .
  * Bleomycine interstitial pneumonitis has been frequently reported and requires the immediate stop of further bleomycine administration.
  * Rarely, procarbazine allergy and intolerance has been reported.
  * Nausea & vomiting due to cyclophosphamide, doxorubicin, dacarbazine and procarbazine may be significant.
  * Total reversible alopecia occurs in most cases.
  * Escalated BEACOPP-related toxic deaths have been reported but do not exceed those observed with standard ABVD.
Long-term toxicity in terms of second malignancies, cardiovascular and pulmonary events | 9 years after FPI

CONTACTS AND LOCATIONS:
Overall Officials: Martin Hutchings, Study Chair — Rigshospitalet, Denmark; Berthe Aleman, Study Chair — The Netherlands Cancer Institute, Amsterdam, The Netherlands; Gustaaf van IMHOFF, Study Chair — University Medical Center Groningen; Wim Oyen, Study Chair — Radboud University Medical Center
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Kreuzberger N, Goldkuhle M, von Tresckow B, Kobe C, Sickinger MT, Monsef I, Skoetz N. Positron emission tomography-adapted therapy for first-line treatment in adults with Hodgkin lymphoma. Cochrane Database Syst Rev. 2025 Mar 26;3(3):CD010533. doi: 10.1002/14651858.CD010533.pub3. PMID 40135712